CLINICAL TRIAL: NCT06908707
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose, Phase 1 Study to Determine the Safety, Tolerability and Pharmacokinetics of LAE102 in Healthy Postmenopausal Women
Brief Title: A Study to Investigate Safety, Tolerability and Pharmacokinetics of LAE102 in Postmenopausal Women
Acronym: LAE102
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laekna Limited (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: LAE102INT1003
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Postmenopausal; Healthy Adult Female Participants
Keywords: Postmenopausal Women

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LAE102 SC (Experimental): Participants will receive a single dose by SC administration (3 dose levels)
  Interventions: Drug: LAE102 SC
- Placebo SC (Placebo Comparator): Participants will receive a single dose by SC administration
  Interventions: Drug: Placebo SC
- LAE102 IV (Experimental): Participants will receive a single IV dose (1 dose level)
  Interventions: Drug: LAE102 IV
- Placebo IV (Placebo Comparator): Participants will receive a single IV dose
  Interventions: Drug: Placebo IV

INTERVENTIONS:
Drug: LAE102 SC — A single dose of LAE102 will be administered subcutaneously
  Other Names: LAE102
  Arms: LAE102 SC
Drug: Placebo SC — A single dose of placebo administered subcutaneously
  Other Names: Placebo
  Arms: Placebo SC
Drug: LAE102 IV — A single dose of LAE102 administered intravenously
  Other Names: LAE102
  Arms: LAE102 IV
Drug: Placebo IV — A single dose of placebo administered intravenously
  Other Names: Placebo
  Arms: Placebo IV

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability and pharmacokinetics (PK) of LAE102 in healthy postmenopausal women

DETAILED DESCRIPTION:
This is a placebo-controlled single ascending dose by subcutaneous (SC) and Intravenous (IV) administration in healthy postmenopausal women to assess the safety and tolerability of LAE102. At least 32 healthy female participants will be enrolled in 4 cohorts with each cohort including 8 participants randomized 6:2 LAE102:Placebo.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 45 to 75 years of age inclusive, at time of signing the informed consent.
* Are healthy postmenopausal female participants.
* Have a body mass index (BMI) within the range 20.0 - 32.0kg/m^2 inclusive at screening.
* Have follicle stimulating hormones (FSH) levels ≥40 IU/L at screening.
* Have clinical laboratory test results within the normal reference range for the population.
* Have venous access sufficient to allow for blood sampling and IV administration of study intervention as per the protocol and have no anticipated contradictions to receiving investigational products via SC administration
* Are capable of giving informed consent.
* Are willing to make themselves available for study visits for the duration of the study and are willing to follow study procedures.

Exclusion Criteria:

* Have a history or presence of clinically significant medical condition(s)
* Have a history of any malignancy within the past 5 years.
* Have hemoglobin level at screening above the upper limit normal for females.
* Have a fasting serum triglyceride level of more than 500mg/dL at screening.
* Have an estimated glomerular filtration rate (eGFR) less than 60mL/min/1.73m^2 at screening.
* Have an abnormal electrocardiogram (ECG)
* Have an abnormal blood pressure.
* Show evidence at screening of HIV or Hepatitis B or C.
* Have a history of or known drug related hypersensitivity or severe allergy
* Underwent major surgery within 30 days prior to study intervention administration or plan to undergo major surgery during the study.
* Have used in the past 90 days or intend to use during the study any medication that may affect FSH levels.
* Have used or intended to use over the counter medications, and/or herbal medicines, from 14 days or 5 half-lives (if known), whichever is longer, prior to study intervention administration until the last visit.
* Received any vaccine 30 days prior to screening or plan to receive any vaccine during the study.
* Have participated, are currently enrolled in, or discontinued from a clinical trial involving an investigational drug or device or off-label use of a drug or device within the last 90 days, or 5-half-lives (if known, whichever is longer), of the last administration of study drug or application of the device, or any other type of medical research judged not to be scientifically or medically compatible with this study.
* Have previously completed or withdrawn from this study or any other study investigating this study intervention.
* Have alcohol consumption exceeding 14 units per week, a positive alcohol test at screening or administration, a history of alcohol abuse within 1 year prior to screening, or are unable to stop alcohol consumption during the study.
* Have a known or suspected history of substance abuse or test positive for drugs of abuse at screening or admission
* Are smoking more than 5 cigarettes (or the equivalent of other tobacco products) per day within 90 days prior to screening or are unable to stop smoking during the study.
* Have donated blood or experienced blood loss of more than 400mL within 90 days prior to screening.
* Are fasting or receiving weight loss treatment within 30 days prior to administration or experiencing major changes in lifestyle.
* In the opinion of the investigator or sponsor and medical monitor, are unsuitable for inclusion in the study.

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Females
Enrollment: 32 (Actual)
Dates: Start 2025-04-22 (Actual); Primary Completion 2025-10-23 (Actual); Study Completion 2025-10-23 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability (number of participants with serious adverse events (SAE)) of LAE102 in healthy postmenopausal women following a single IV or SC dose | Baseline up to 8 weeks
  Number of participants with SAEs
  - Evaluation of Safety and Tolerability of LAE102
To evaluate the safety and tolerability (number of participants with treatment emergent adverse events (TEAE)) of LAE102 in healthy postmenopausal women following a single IV or SC dose | Baseline up to 8 weeks
  Number of participants with TEAEs
  - Evaluation of Safety and Tolerability of LAE102

SECONDARY OUTCOMES:
To evaluate the Maximum Concentration (Cmax) of LAE102 in healthy postmenopausal women following a single IV or SC dose | Predose up to 8 weeks
  - PK: Cmax of LAE102
To evaluate the Area Under Curve (AUC) of LAE102 in healthy postmenopausal women following a single IV or SC dose | Predose up to 8 weeks
  - PK: AUC of LAE102
To evaluate the Time of Maximum Serum Concentration (Tmax) of LAE102 in healthy postmenopausal women following a single IV or SC dose | Predose up to 8 weeks
  - PK: Tmax of LAE102

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Hugh Coleman, MD, Principal Investigator — Fortrea Clinical Research Unit Inc.
Locations (1):
- Fortrea Clinical Trials, Daytona Beach, Florida, United States